CLINICAL TRIAL: NCT01954732
Title: A Pharmacodynamic Study of Metformin in Patients With Resectable Pancreatic Cancer
Brief Title: Metformin Hydrochloride in Treating Patients With Pancreatic Cancer That Can be Removed by Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE1213; NCI-2013-01836 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 1213 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (observation) (No Intervention): Patients undergo observation.
- Group II (metformin hydrochloride) (Experimental): Patients receive metformin hydrochloride PO BID for at least 7 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: metformin hydrochloride; Other: pharmacological study
- Group III (metformin hydrochloride) (Experimental): Patients receive metformin hydrochloride as in Group II.
  Interventions: Drug: metformin hydrochloride; Other: pharmacological study

INTERVENTIONS:
Drug: metformin hydrochloride — Given PO
  Other Names: Glucophage
  Arms: Group II (metformin hydrochloride); Group III (metformin hydrochloride)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
  Arms: Group II (metformin hydrochloride); Group III (metformin hydrochloride)

SUMMARY:
This randomized clinical trial studies metformin hydrochloride in treating patients with pancreatic cancer that can be removed by surgery. Metformin hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of escalating doses of metformin (metformin hydrochloride) given pre-operatively on pancreatic cancer cell proliferation and apoptosis.

SECONDARY OBJECTIVES:

I. To assess toxicity of escalating doses of metformin given pre-operatively in patients with resectable pancreatic carcinoma.

II. To measure the effect of metformin on the expression of phosphorylated acetyl-CoA carboxylase alpha (ACC), phosphorylated mechanistic target of rapamycin (serine/threonine kinase) (mTOR), and pancreatic cancer stem cells.

OUTLINE: Patients are randomized to 1 of 3 treatment groups.

GROUP I: Patients undergo observation.

GROUP II: Patients receive metformin hydrochloride orally (PO) twice daily (BID) for at least 7 days in the absence of disease progression or unacceptable toxicity.

GROUP III: Patients receive metformin hydrochloride as in Group II.

After completion of study treatment, patients are followed up 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed resectable pancreatic carcinoma; patients with pancreatic neuroendocrine tumors are not eligible
* Patients must be previously untreated with chemotherapy or radiation therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must have surgical resection of the pancreas planned, with enrollment at least 7 days prior to surgery; patients with surgery scheduled > 15 days will not be excluded
* Hemoglobin (Hg)A1C must be below 7%
* Total bilirubin less than 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 X institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Serum creatinine within normal institutional limits
* Alkaline phosphatase < 1.5 X institutional upper limit of normal
* Subjects must have the ability to understand and be willing to provide written informed consent

Exclusion Criteria:

* History of metformin use in the previous 3 months
* Treatment with neoadjuvant chemotherapy or radiation therapy
* History of allergic reactions attributed to metformin
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Metabolic acidosis, acute or chronic, including ketoacidosis
* Metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pancreatic tumor cell proliferation and apoptosis as measured by the percentage of cells Ki-67+, percentage of cells TUNEL+, and mitotic counts in tissue samples | At time of surgery (after 7 days of treatment)
  The difference between treatment groups will be compared using analysis of variance (ANOVA) (3 groups) followed by Tukey's pair-wise comparison procedure. Transformation may be applied (e.g. natural log) prior to analysis to better approximate normality.

SECONDARY OUTCOMES:
Occurrence of grade 3 and 4 toxicities according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE; version 4.0) | Baseline to 30 days after treatment has been discontinued or after the date of surgery, whichever occurs first
  Will be summarized as the percentage of patients by type and grade according to treatment group.
Expression of pACC and pMTOR quantified by the mean fluorescence intensity (MFI) in tissue samples | At time of surgery (after 7 days of treatment)
  The difference between treatment groups will be compared using ANOVA followed by Tukey's pair-wise comparison procedure. Laser scanning cytometry and iCyte software used to quantify the MFI of pACC and pMTOR.
Percentage of pancreatic cancer stem cells in tissue samples | At time of surgery (after 7 days of treatment)
  For each of biologic biomarkers (pACC, pMTOR, CD44+CD24+ESA+ cells), the difference between treatment groups will be compared using ANOVA (3 groups) followed by Tukey's pair-wise comparison procedure. Transformation may be applied (e.g. natural log) prior to analysis to better approximate normality.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Eads, MD, Principal Investigator — Case Comprehensive Cancer Center